CLINICAL TRIAL: NCT02796586
Title: Salt Lake Refugee Women's Health Project-Group Versus Individual Contraceptive Counseling for Resettled African Refugee Women
Brief Title: Group Versus Individual Contraceptive Counseling for Resettled African Refugee Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Par Royer, Adjunct Faculty, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00080655
Record Dates: First submitted 2016-05-13; First posted 2016-06-10 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Contraception
Keywords: Refugee Health; Resettled Refugee; Family Planning; Contraception; Group Counseling; Group contraceptive counseling
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual Contraceptive Counseling (Placebo Comparator): Performed by a medical provider and planned to simulate a typical clinic visit addressing contraception.
  Interventions: Other: Counseling
- Group Contraceptive Counseling (Experimental): Performed by a bicultural study staff member who speaks the primary languages of participants and had been formally trained in contraception counseling.
  Interventions: Other: Counseling

INTERVENTIONS:
Other: Counseling — Participants will be randomly assigned to group versus individual contraceptive counseling

SUMMARY:
To evaluate the feasibility and effectiveness of group contraceptive counseling on family planning knowledge acquisition, service satisfaction, method uptake and continuation among a group of resettled African refugee women.

DETAILED DESCRIPTION:
Thousands of women refugees arrive in the United States each year, yet there is very little known about reproductive health and family planning needs of these women after resettlement.

This randomized controlled pilot study, in a population of resettled African refugee women, will evaluate differences between group and individual contraceptive counseling on the decision to use contraception, satisfaction with counseling method, and modern family planning knowledge.

Participants will arrive to clinic during an assigned "intervention day." An intake and exit survey will be performed before and after their counseling session. Demographics, attitudes towards contraception, and knowledge regarding contraceptive methods will be assessed via questionnaire. Participants will be randomized to either group or individual contraceptive counseling. After each session, participants will have the option to privately choose a reversible method of contraception free of charge.

Telephone survey follow-up with participants will occur every three months for one year. Follow-up surveys will include questions regarding method continuation, method satisfaction and and modern contraceptive knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Resettled refugee
* Ability to speak and comprehend conversational Swahili, French or Lingala
* Interest in contraceptive counseling
* Willing to adhere to study protocols including randomization and follow-up
* Cellular phone access

Exclusion Criteria:

* Male

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Knowledge Acquisition assessed via number of correct questions on modified FogZone questionnaire | Day of intervention (Study Day 1)
  Evaluate knowledge acquisition by comparing results on pre and post test of modern contraceptive knowledge. Contraceptive knowledge will be assessed using a modified version of the FogZone questionnaire
Contraceptive uptake | Day of intervention (Study day 1)
  Evaluate contraceptive uptake via query of method choice after counseling
Service Satisfaction via questionnaire | Day of intervention (Study day 1)
  Evaluate satisfaction with service and type of counseling received using questionnaire
Service satisfaction via Likert Scale | Day of intervention (Study day 1)
  Evaluate satisfaction with service and type of counseling received using questionnaire

SECONDARY OUTCOMES:
Method Continuation | 3, 6, 9 and 12 months post-intervention
  Evaluate method continuation via telephone survey
Knowledge Retention assessed via modified FogZone questionnaire | 3, 6, 9 and 12 months post-intervention
  Evaluate knowledge retention by repeating knowledge questionnaire and comparing baseline and interval results.

CONTACTS AND LOCATIONS:
Overall Officials: Par Royer, MD MSCI, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No